CLINICAL TRIAL: NCT03979430
Title: Early Detection of Acute Exacerbation in Patients With Idiopathic Lung Fibrosis - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: University of Giessen (Other); Hannover Medical School (Other); Ludwig-Maximilians - University of Munich (Other); LungenClinic Grosshansdorf (Other)
Responsible Party: Principal Investigator, Michael Kreuter, Principal Investigator, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AE-IPF study
Record Dates: First submitted 2019-05-14; First posted 2019-06-07 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Acute Exacerbation; Idiopathic Pulmonary Fibrosis; Home Spirometry
Keywords: Acute Exacerbation; Idiopathic Pulmonary Fibrosis; Home Spirometry
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Intervention group on 5 different sites without a control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): There is only one arm with the intervention.
  Interventions: Other: Home spirometry

INTERVENTIONS:
Other: Home spirometry — Patients will receive a tablet and a spirometer for daily home spirometry. Each patient is supposed to do the home spirometry at the same time every morning. The spirometer and the tablet are connected via Bluetooth. Data will be transferred to a webpage, which team members have access to. Alerts will be automatically send to team members, if the FVC-value decreases about 5% or more within three consecutive days or if the patient does not do the measurement on three consecutive days. Study period is one year. Patients will also conduct a survey to measure health related quality of life (K-BILD). This questionnaire, as well as a phone interview to record changes in medication and condition will be conducted at baseline and every 4 weeks. At baseline and after 3, 6, 9, and 12 months, patients will conduct a 6 minutes walking test, lung function test, blood will be drawn for biomarker analysis, and sputum, nasal swab, and urine samples will be collected and analyzed.

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a chronic disease, leading to poor lung function with a median survival of 2-3 years. Acute exacerbation of idiopathic IPF is a complication associated with a mortality rate > 50%. So far, the appearance of an acute exacerbation is unpredictable. Worsening of the IPF accompanies with a decrease of the FVC-value, the lung capacity. So far, studies are missing investigating the correlation between a decrease of the FVC-value and emerging acute exacerbations. Therefore, this study uses daily home spirometry to investigate that correlation. With this study the investigators hope to determine acute exacerbations early and treat patients early.

DETAILED DESCRIPTION:
This study is a multi-Center study happening on five different sites, Heidelberg, Gießen, Grosshansdorf, München, and Hannover, all in Germany. Each site recuits ten patients for a total of 50 patients.

All patients will receive a tablet and a spirometer for daily home spirometry. Each patient is supposed to do the home spirometry at the same time every morning. The spirometer and the tablet are connected via Bluetooth and data will be transferred to a webpage after the measurement, that team members have access to the data and can see the progress daily. Alerts will be automatically send to team members, if the FVC-value decreases about 5% or more within three consecutive days or if the patient does not do the measurement on three consecutive days. Study period is one year.

In addition to the home spirometry, patients will conduct a survey to measure health related quality of life (K-BILD). This questionnaire will be conducted at baseline and then every 12 weeks. Every 4 weeks the patients are participating in a phone interview to record changes in medication and condition. At baseline and after 3, 6, 9, and 12 months, patients will conduct a 6 minutes walking test, lung function test, blood will be drawn for biomarker analysis, and sputum, nasal swab, and a urine sample will be collected and analyzed.

Aim is to detect and treat an acute exacerbation early.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the study
* diagnosis of IPF
* Age > 18 years
* FVC < 70%
* DLCO-SB <60%
* Ability to work with a tablet and home spirometer

Exclusion Criteria:

* Patient does not understand the study
* Patient cannot participate in study related processes
* pulmonary infection within the last 4 weeks
* acute exacerbation within the last 4 weeks
* obstructive Ventilation disorders
* other respiratory decline within the last 4 weeks
* relevant malignancy within the last 5 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation of change in FVC-values and the appearance of an acute exacerbation | Each participant will be followed for one year
  A decrease in FVC value can predict an acute exacerbation. Through daily home spirometry, study team members have access to measured FVC-values from each patient. Therefore, changes in FVC values can be seen directly and actions can be taken to detect an acute exacerbation or even to avoid one.

SECONDARY OUTCOMES:
Correlation between spirometry and early detection of an acute exacerbation | 1 year
  Identifying an acute exacerbation early is important for further treatment of ILD patients. With home spirometry, the investigators want to examine the feasibility of such measurements.
Correlation between home spirometry and health related quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kreuter, Prof., Principal Investigator — Heidelberg University
Locations (4):
- Germany (4):
  - University of Gießen-Marburg, Giessen
  - LungenClinic Grosshansdorf, Großhansdorf
  - Medical University Hannover, Hanover
  - CPC Comprehensive Pneumology Center, München

IPD SHARING:
Plan to Share IPD: No